CLINICAL TRIAL: NCT06959199
Title: EndoVascular Treatment Beyond 24 Hours for AcutE Ischemic Stroke Caused by Anterior Circulation LArge Vessel STEnosis: A Multicenter RandomizeD Controlled Trial(EVT-BELATED)
Brief Title: Endovascular Treatment Beyond 24 Hours for Acute Ischemic Stroke Caused by Anterior Circulation Large Vessel Stenosis
Acronym: EVT-BELATED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Qi Li, Professor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YX2024-241(F1)
Record Dates: First submitted 2025-04-26; First posted 2025-05-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Ischemic Stroke; Infarction
Keywords: Ischemic stroke; Endovascular therapy; Stroke
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Ischemic Stroke; Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Treatment plus Best Medical Treatment (Experimental): Patients in this group will receive endovascular therapy (EVT) plus best medical treatment.
  Interventions: Procedure: Endovascular Treatment; Drug: Best Medical Treatment
- Best Medical Treatment (Active Comparator): Patients in this group will receive standard medical therapy in accordance with the guideline-directed management for acute ischemic stroke.
  Interventions: Drug: Best Medical Treatment

INTERVENTIONS:
Procedure: Endovascular Treatment — EVT procedures may include mechanical thrombectomy, intra-arterial thrombolysis, balloon angioplasty, or stenting, or other intra-arterial procedures as deemed appropriate by the treating physician.
  Arms: Endovascular Treatment plus Best Medical Treatment
Drug: Best Medical Treatment — Patients in this group will receive standard medical therapy in accordance with the guideline-directed management for acute ischemic stroke.

SUMMARY:
Endovascular therapy (EVT) is currently recommended as the first-line treatment for patients with acute large vessel occlusion (LVO) in the anterior circulation within 24 hours of symptom onset. However, the therapeutic benefit of EVT beyond 24-hour window remains uncertain due to limited evidence. The EVT-BELATED trial is a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) study designed to assess the safety and efficacy of EVT in patients with acute ischemic stroke (AIS) caused by anterior circulation LVO presenting beyond 24 hours after symptom onset.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) trial. Eligible participants will be adults (age >18 years) presenting with acute ischemic stroke (AIS) due to anterior circulation large vessel occlusion (LVO), either with a time window of 24 to 120 hours from symptom onset or last known well or progressive ischemic stroke with a time from symptom onset of 24 hours to 7 days. Participants who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned in a 1:1 ratio to one of two treatment arms. The control group will receive best medical management alone, while the intervention group will receive best medical management in combination with endovascular therapy (EVT). EVT procedures may include mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty, or stenting, as deemed appropriate by the treating physician.

The primary objective of the study is to evaluate the safety and efficacy of EVT in patients presenting with AIS due to anterior circulation LVO beyond 24 hours from symptom onset. The primary endpoint is functional independence at 90 days, defined as a score of 0-2 on the modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Acute ischemic stroke with a time window of 24 to 120 hours from symptom onset or last known well, or progressive ischemic stroke with a time from symptom onset of 24 hours to 7 days (A ≥4-point increase in NIHSS attributable to the culprit vessel territory )
* NIHSS score 5-25
* Occlusion or ≥70% stenosis of the internal carotid artery or the M1/M2 segment of the middle cerebral artery, confirmed by CTA, MRA, or DSA, and deemed to be the culprit vessel responsible for the clinical presentation of acute ischemic stroke
* Meet one of the following imaging criteria:

  1. MRI-based criteria: the infarct volume on DWI is less than one-third of the MCA territory, with evidence of DWI-FLAIR mismatch or MR perfusion showing a core infarct volume ≤30 ml, a mismatch ratio ≥1.8, and a mismatch volume ≥15 ml;
  2. CTA-based criteria: good collateral circulation on the affected side defined ascollateral filling >50% of the MCA territory (Tan score ≥2) and an ASPECTS score ≥6);
  3. CTP-based criteria: ischemic core volume ≤30 ml, mismatch ratio ≥ 1.8, and mismatch volume ≥ 15mL
* Signed informed consent obtained

Exclusion criteria:

* Pre-stroke mRS ≥ 2
* Patients unable to undergo vascular imaging
* Patients with known allergies to iodine contrast agents, anesthetics, or any contraindication to endovascular treatment
* Prior endovascular therapy performed after the index stroke event during the current hospitalization
* Intracranial hemorrhage identified on initial imaging
* Platelet count <50×10⁹/L, or presence of a known hemorrhagic diathesis , coagulation factor deficiencies, or use of oral anticoagulation therapy with an International Normalized Ratio (INR) > 3.0
* Refractory hypertension, defined as sustained systolic blood pressure >200 mmHg or diastolic blood pressure >120 mmHg despite optimal medical management
* History of intracranial hemorrhage within the past 3 months, including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, epidural hemorrhage, or subdural hemorrhage
* Significant mass effect with midline shift confirmed by CT or MRI
* Suspected cardioembolic stroke or stroke due to non-atherosclerotic etiologies, such as:arterial dissection,Moyamoya disease, Infective endocarditis, or Immune-mediated vasculitis
* Prior intracranial stent placement in the same culprit vessel
* Major surgery performed within the past 30 days
* Pregnant or current breastfeeding
* Presence of severe systemic comorbidities with a life expectancy of less than 3 months
* Deemed unsuitable for participation by the investigator for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional independence | 90 ± 7 days
  The proportion of patients achieving functional independence, defined as a modified Rankin Scale (mRS) score of 0-2 at 90 ± 7 days.
  The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Ordinal distribution of mRS | 90 ± 7 days
  Ordinal distribution of the modified Rankin Scale (mRS) at 90 ± 7 days. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Excellent functional outcome | 90 ± 7 days
  Number of participants achieving an excellent functional outcome, defined as a modified Rankin Scale (mRS) score of 0-1 at 90 ± 7 days follow-up. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Poor functional outcome | 90 ± 7 days
  Number of participants achieving a poor functional outcome, defined as a modified Rankin Scale (mRS) score of 4-6 at 90 ± 7 days follow-up. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Early neurological deterioration | 24 ± 12 hours
  The proportion of patients with an increase of ≥ 4 points in the National Institutes of Health Stroke Scale (NIHSS) score, within 24 ± 12 hours post-randomization. The NIHSS is a standardized 11-item assessment tool designed to quantify neurological deficits in patients with acute stroke. The total score ranges from 0 to 42, with higher values indicating more severe deficits.
Any neurological improvement | 24 ± 12 hours
  The proportion of patients with a reduction of ≥ 2 points in the National Institutes of Health Stroke Scale (NIHSS) score from baseline at 24 ± 12 hours post-randomization. The NIHSS is a standardized 11-item assessment tool designed to quantify neurological deficits in patients with acute stroke. The total score ranges from 0 to 42, with higher values indicating more severe deficits.
Early neurological improvement | 24 ± 12 hours
  The proportion of patients with a reduction of ≥ 4 points in the National Institutes of Health Stroke Scale (NIHSS) score from baseline at 24 ± 12 hours post-randomization. The NIHSS is a standardized 11-item assessment tool designed to quantify neurological deficits in patients with acute stroke. The total score ranges from 0 to 42, with higher values indicating more severe deficits.
Any new ischemic stroke events | 3 months
  Any new ischemic stroke events within 3 months
Any ischemic stroke event or revascularization | 3-12 months
  Any ischemic stroke event or revascularization of the culprit vessel between 3 and 12 months post-randomization.

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage | 24 ± 12 hours
  The incidence of symptomatic intracranial hemorrhage within 24 ± 12 hours post-randomization.
All cause mortality | 90 ± 7 days
  All cause mortality at 90 ± 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second (Affiliated) Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided